CLINICAL TRIAL: NCT04320134
Title: CliNIcal SCEnarios and Pathophysiological Features of Patients With Atrial Fibrillation: a Long Term Prospective Study (NICE-AF Study)
Brief Title: cliNIcal sCEnarios and Pathophysiology of Atrial Fibrillation
Acronym: NICE-AF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, Professor, FESC, Policlinico Casilino ASL RMB
Other Study IDs: PoliclinicoCasilino1-2020
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pathophysiology; triggers; substrates; autonomic system
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation (AF) remains the most common sustained cardiac arrhythmia with prevalence and incidence continuously increasing worldwide. Current guidelines propose an etiological, symptom-based classification of the arrhythmia and mainly focused on its duration with consequent rhythm or rate-control strategies. Moreover, risk scores for atherothrombotic systemic or hemorrhagic events related to atrial fibrillation are principally based on patients cardiovascular history and risk factors.

This approach do not consider relevant pathophysiological aspects that may play a pivotal role in triggering or perpetuating the arrhythmia, especially at its first occurrence. At this point, a crucial step would be deeply investigating AF clinical and pathophysiological features to guide a tailored diagnostical and therapeutic approach. Indeed, early recognition and proper characterization of triggers, substrates, autonomic system imbalance and modulating factors (drugs, electrolytes, etc) are of the utmost importance for AF care and management.

Therefore, this large scale prospective observational study aims to evaluate clinical and pathophysiological features of patients with symptomatic and asymptomatic atrial fibrillation in different scenarios to understand possible distinctive characteristics warranting a personalized approach to the arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with electrocardiographic diagnosis of Atrial Fibrillation (New Onset, Paroxysmal, Persistent, Long Standing Persistent and Permanent) admitted to the Emergency Room and/or Cardiology Department /ambulatory care center of our Hospital
* Age >18 years old
* Patients who can give their written informed consent.

Exclusion Criteria:

* Age <18 years old
* Patients who cannot give their written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective observational study we consider to enroll patients with diagnosis of Atrial Fibrillation (new onset, paroxysmal, persistent, long-persistent and permanent) admitted to our Hospital in the Emergency Room and/or Cardiology Department/Ambulatory Care Center.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Atrial Fibrillation recurrences | 5 years
  frequency distribution
Number of participants with Major Adverse Cardiac Events (MACE) | 5 years
  frequency distribution
Rate of thromboembolic events | 5 years
  frequency distribution
Rate of bleeding events | 5 years
  frequency distribution of minor, major and fatal bleedings

SECONDARY OUTCOMES:
Rate of participants socio-demographic characteristics | baseline and 5 years
  Frequency distribution: age, gender, race, occupation, life-style, diet, physical activity, alcohol consumption
Rate of participants with comorbidities | baseline and 5 years
  Frequency distribution: hypertension, heart failure, diabetes mellitus, kidney failure, dyslipidemia, lung diseases, thyroid disorders, gastrointestinal and liver disorders, hematological diseases, neoplasms, autoimmune disorders
Rate of participants with Heart diseases | baseline and 5 years
  frequency distribution: vascular diseases, valvular problems, cardiomyopathies, arrhythmias, family/genetic history of cardiovascular disease
Rate of patients with Atrial Fibrillation secondary to triggers and/or autonomic system imbalance and/or modifiable factors | baseline and 5 years
  Frequency distribution of patients in which atrial fibrillation was clearly related to adrenergic tone imbalance and/or vagal tone imbalance and/or secondary to modifiable factors
Describe imaging parameters (echocardiogram and cardiac magnetic resonance) | baseline and 5 years
  Left ventricle, right ventricle, right and left atrium and valves: morphologies, volumes, dimensions and function
Concentration of laboratory biomarkers | baseline and 5 years
  Complete Blood cell count with differential; Interleukin-1, Interleukin-6, High sensitivity C Reactive protein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curtis AB, Gersh BJ, Corley SD, DiMarco JP, Domanski MJ, Geller N, Greene HL, Kellen JC, Mickel M, Nelson JD, Rosenberg Y, Schron E, Shemanski L, Waldo AL, Wyse DG; AFFIRM Investigators. Clinical factors that influence response to treatment strategies in atrial fibrillation: the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Am Heart J. 2005 Apr;149(4):645-9. doi: 10.1016/j.ahj.2004.09.038. PMID 15990747
- [Background] Siontis KC, Gersh BJ, Killian JM, Noseworthy PA, McCabe P, Weston SA, Roger VL, Chamberlain AM. Typical, atypical, and asymptomatic presentations of new-onset atrial fibrillation in the community: Characteristics and prognostic implications. Heart Rhythm. 2016 Jul;13(7):1418-24. doi: 10.1016/j.hrthm.2016.03.003. Epub 2016 Mar 4. PMID 26961300
- [Background] Heijman J, Guichard JB, Dobrev D, Nattel S. Translational Challenges in Atrial Fibrillation. Circ Res. 2018 Mar 2;122(5):752-773. doi: 10.1161/CIRCRESAHA.117.311081. PMID 29496798
- [Background] Rienstra M, Vermond RA, Crijns HJ, Tijssen JG, Van Gelder IC; RACE Investigators. Asymptomatic persistent atrial fibrillation and outcome: results of the RACE study. Heart Rhythm. 2014 Jun;11(6):939-45. doi: 10.1016/j.hrthm.2014.03.016. Epub 2014 Mar 13. PMID 24632222
- [Background] Frykman V, Frick M, Jensen-Urstad M, Ostergren J, Rosenqvist M. Asymptomatic versus symptomatic persistent atrial fibrillation: clinical and noninvasive characteristics. J Intern Med. 2001 Nov;250(5):390-7. doi: 10.1046/j.1365-2796.2001.00893.x. PMID 11887973
- [Background] Chung MK, Eckhardt LL, Chen LY, Ahmed HM, Gopinathannair R, Joglar JA, Noseworthy PA, Pack QR, Sanders P, Trulock KM; American Heart Association Electrocardiography and Arrhythmias Committee and Exercise, Cardiac Rehabilitation, and Secondary Prevention Committee of the Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; and Council on Lifestyle and Cardiometabolic Health. Lifestyle and Risk Factor Modification for Reduction of Atrial Fibrillation: A Scientific Statement From the American Heart Association. Circulation. 2020 Apr 21;141(16):e750-e772. doi: 10.1161/CIR.0000000000000748. Epub 2020 Mar 9. PMID 32148086
- [Background] Slomski A. Alcohol Abstinence Lowers Atrial Fibrillation Recurrence Risk. JAMA. 2020 Feb 25;323(8):701. doi: 10.1001/jama.2020.1005. No abstract available. PMID 32096848
- [Background] Stiell IG, Sivilotti MLA, Taljaard M, Birnie D, Vadeboncoeur A, Hohl CM, McRae AD, Rowe BH, Brison RJ, Thiruganasambandamoorthy V, Macle L, Borgundvaag B, Morris J, Mercier E, Clement CM, Brinkhurst J, Sheehan C, Brown E, Nemnom MJ, Wells GA, Perry JJ. Electrical versus pharmacological cardioversion for emergency department patients with acute atrial fibrillation (RAFF2): a partial factorial randomised trial. Lancet. 2020 Feb 1;395(10221):339-349. doi: 10.1016/S0140-6736(19)32994-0. PMID 32007169